CLINICAL TRIAL: NCT02299401
Title: Assessing the Effectiveness of Two Regimens of Misoprostol Alone for Early Pregnancy Termination and Use of a Semi-Quantitative Pregnancy Test for At-Home Follow-Up
Brief Title: Effectiveness of Two Regimens of Misoprostol Alone for Early Pregnancy Termination and Use of SQPT for At-Home Follow-Up
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6006
Record Dates: First submitted 2014-11-13; First posted 2014-11-24 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Pregnancy
Keywords: Medical abortion; Induced abortion; Pregnancy test; Semi-quantitative pregnancy test
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buccal (Experimental): Women randomized to receive three 800 mcg doses of misoprostol taken buccally in three hour intervals. All women receive a semi-quantitative pregnancy test for at-home follow up.
  Interventions: Drug: Misoprostol; Device: Semi-quantitative pregnancy test
- Sublingual (Experimental): Women randomized to receive three 800 mcg doses of misoprostol taken sublingually in three hour intervals. All women receive a semi-quantitative pregnancy test for at-home follow up.
  Interventions: Drug: Misoprostol; Device: Semi-quantitative pregnancy test

INTERVENTIONS:
Drug: Misoprostol — Women will receive three 800 mcg doses of misoprostol.
Device: Semi-quantitative pregnancy test — All women will be given a semi-quantitative pregnancy test (SQPT) for at-home follow-up.
  Other Names: SQPT

SUMMARY:
This randomized trial will compare the rates of ongoing pregnancy, safety/side effects and acceptability of two medical abortion regimens that are commonly used in Latin America. The first regimen will involve three 800 mcg doses of misoprostol taken buccally in three hour intervals; the second will involve three 800 mcg doses of misoprostol taken sublingually in three hour intervals. This study will also aim to assess the feasibility and acceptability of a semi-quantitative pregnancy test (SQPT) for at-home follow-up in both settings.

ELIGIBILITY:
Inclusion Criteria:

* Presents for voluntary termination of pregnancy
* Gestational age ≤ 70 days by last menstrual period plus clinical assessment or ultrasound
* General good health including the absence of conditions which contraindicate the use of misoprostol for pregnancy termination
* Agrees to return for follow-up visit and willing to provide an address and/or telephone number for the purposes of follow-up
* Able to consent to study participation

Exclusion Criteria:

* Gestational age > 70 days last menstrual period
* Confirmed or suspected ectopic or molar pregnancy
* Contraindications to medical abortion include having an intrauterine device in place and history of allergy to misoprostol or other prostaglandins

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2014-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rates | 1-2 weeks
  The study will assess and compare the rates of ongoing pregnancy for the two medical abortion regimens at 1-2 week follow up.

SECONDARY OUTCOMES:
Incidence of side effects and complications as a measure of safety/ side effects | 1-2 weeks
  Assess and compare the safety/side effects of two regimens of misoprostol alone for early pregnancy termination.
Reported acceptability and satisfaction with misoprostol regimen | 1-2 weeks
  The study will also assess and compare satisfaction and acceptability of each medical abortion regimen as rated by the women.
Usability of SQPT as measured by women's ability to assess success of medical abortion procedure at home | 1-2 weeks
  The study will assess women's ability to use the SQPT effectively for at-home assessment of the success of the medical abortion procedure.
Self-reported acceptability and satisfaction with SQPT as a means of at-home follow up | 1-2 weeks
  The study will also assess the acceptability of the test as a means for at-home follow-up after medical abortion as rated by the women. The woman will answer questions about whether she found the SQPT easy to use an acceptable for at-home follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy R Sheldon, PhD, Study Director — Gynuity Health Projects
Locations (2):
- Reproductive Health Clinic, La Paz, Pedro Domingo Murillo, Bolivia
- Reproductive Health Clinic, Quito, Ecuador

REFERENCES:
- [Derived] Sheldon WR, Durocher J, Dzuba IG, Sayette H, Martin R, Velasco MC, Winikoff B. Early abortion with buccal versus sublingual misoprostol alone: a multicenter, randomized trial. Contraception. 2019 May;99(5):272-277. doi: 10.1016/j.contraception.2019.02.002. Epub 2019 Mar 1. PMID 30831103